CLINICAL TRIAL: NCT05685316
Title: Pilot Clinical Trial to Evaluate the Preliminary Safety and Performance of COPLA® for Treatment of Cartilage Defects
Brief Title: COPLA® Cartilage Implant Pilot Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Askel Healthcare Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU06-001
Record Dates: First submitted 2022-12-19; First posted 2023-01-17 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cartilage or Osteochondral Defects in the Knee
Keywords: Cartilage; Cartilage lesion; Cartilage defect; Knee cartilage; Cartilage repair; Chondral defect; Osteochondral defect

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPLA® cartilage implant (Experimental): The potential subjects will be screened against inclusion and exclusion criteria. If deemed eligible, they will be consented and enrolled. The enrolled subjects will receive COPLA® device during normal clinical practice for cartilage repair surgery with bone marrow stimulation.
  Interventions: Device: COPLA® cartilage implant

INTERVENTIONS:
Device: COPLA® cartilage implant — In the investigation, the subjects will receive COPLA® device during normal clinical practice for cartilage repair surgery of the knee with bone marrow stimulation.

SUMMARY:
This is a first-in-human clinical, open label, non-randomized, prospective investigation to assess the initial safety and performance of the COPLA® cartilage implant. In the investigation, the patients will receive COPLA® device during normal clinical practice for cartilage repair surgery with bone marrow stimulation.

DETAILED DESCRIPTION:
Included subjects will be symptomatic patients between the ages 18 and 50 years with a single contained chondral or osteochondral defect located on the femoral condyle and graded as III or IV according to the International Cartilage Repair Society (ICRS) grading system. Subjects with known health related risks or certain recent surgical or medical interventions will be excluded.

The primary objective of the investigation is to confirm that COPLA® device is safe for humans. The secondary objectives relate to the performance of the device after it is placed into the knee joint during surgery. Focus points of secondary objectives will be facilitation of mobility and non-restricted weight-bearing of the operated leg as well as the identification of repair tissue growth at the lesion site.

Post-operative follow-up is planned for 24 months after surgery. Subject will come for scheduled visits at 6-week, 3-month, 6-month, 12-month, and 24-month timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Single contained symptomatic chondral or osteochondral defect located on the femoral condyle graded as ICRS III or IV observed in the preoperative MRI;
2. Minimum defect size 1 cm2 post-debridement;
3. Aged between 18 and 50 at the time of enrollment;
4. Osteoarthritis of the index knee graded 0 or I according to the Kellgren-Lawrence Grading in posterior-anterior knee radiography with full weight bearing;
5. Subject is able and willing to give informed consent; AND
6. Subject is physically and mentally willing and able to comply with the post-operative rehabilitation protocol, questionnaires, and scheduled clinical and radiographic visits

Exclusion Criteria:

1. Defect size over 4 cm2 according to arthroscopy during operation;
2. Subchondral defect depth over 4 mm according to pre-operative MRI;
3. Osteoarthritis of the index knee grades II or above according to the Kellgren-Lawrence Grading;
4. History of allergic reaction or intolerance of materials containing polylactide and/or bovine collagen;
5. Presence of an additional articular cartilage lesions in the femur, tibia or the patella, ICRS grades III or above observed in the preoperative MRI or during the final intraoperative arthroscopic evaluation;
6. Any known systemic cartilage and/or bone disorder, such as but not limited to, osteochondrosis, osteoporosis, chondrodysplasia or osteogenesis imperfecta;
7. Any previous surgical treatment in the index knee in the past 12 months;
8. Any previous intra-articular injections in the index knee in the past 3 months;
9. Systemic corticosteroid therapy in the past 1 month;
10. Presence of an untreated clinically significant meniscal tear;
11. Lack of functional remaining meniscus, at least 5mm rim at the end of the procedure;
12. Prior meniscal resection > 50%;
13. Untreated Anterior cruciate ligament (ACL) and/or Posterior cruciate ligament (PCL) deficiency: collateral and rotational;
14. Anteroposterior and/or varus/valgus instability on clinical testing;
15. Asymmetrical collateral stability in full extension and 20-degree flexion on clinical testing;
16. Need for any concomitant surgical intervention with the cartilage repair;
17. Inflammatory joint disease of the index or contralateral knee;
18. Any known history of inflammatory arthropathy or crystal-deposition arthropathy;
19. Active acute or chronic intra-articular or osseous infection of the index knee;
20. Any evidence of active infection anywhere in the body;
21. Inflammatory joint disease;
22. Body Mass Index (BMI) ≥ 30;
23. History of any significant systemic disease, such as but not limited to: human immunodeficiency virus (HIV), hepatitis, human T-lymphotropic virus (HTLV), syphilis, and coagulopathies;
24. Use of anticoagulation medication or antiaggregant medication; however up to 100 mg Acetylsalicylic acid (ASA) daily is allowed;
25. Chemotherapy in the past 12 months;
26. Any known tumor of the index knee;
27. Subject known to be pregnant or lactating;
28. Participation in other clinical trials within 60 days prior to this trial or concurrent with this trial;
29. Prisoners;
30. Known substance or alcohol abuse; OR
31. Current nicotine users

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of Serious Adverse Events (SAE) | From pre-operative baseline up to 24-month follow-up visit
  Safety - Measured by number of SAE and evaluated over the course of the clinical investigation

SECONDARY OUTCOMES:
Defect filling | From pre-operative baseline up to 24-month follow-up visit
  Measured by the change in repair tissue quality evaluated according to Magnetic Resonance Imaging (MRI) Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART 2.0)
Change in pain score | From pre-operative baseline up to 24-month follow-up visit
  Measured by the change in pain score according to the Knee Injury and Osteoarthritis Outcome Score (KOOS) pain subscale (scale from never to always).
Functional outcome | From pre-operative baseline up to 24-month follow-up visit
  Measured by the change in joint function scores according to the KOOS joint function subscales (degree of difficulty, scale from none to extreme).
Change in Quality of life | From pre-operative baseline up to 24-month follow-up visit
  Measured by the change to 12-Item Short Form Survey (SF-12) Health Survey (scale from excellent to poor).

CONTACTS AND LOCATIONS:
Locations (6):
- Tartu University Hospital, Tartu, Estonia
- Finland (4):
  - Mehiläinen, Helsinki
  - Terveystalo, Helsinki
  - Central Finland Health Care District, Jyväskylä
  - Terveystalo, Jyväskylä
- Sahlgrenska University hospital, Gothenburg, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No